CLINICAL TRIAL: NCT05090683
Title: Evaluation of a Mind-body Based Application for the Treatment of Chronic/Persistent Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Fraser Valley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100820
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-12

CONDITIONS: Chronic Pain; Migraine; Chronic Pain Syndrome
Keywords: chronic pain; mind-body; mobile application
MeSH Terms: conditions — Chronic Pain; Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two groups: control (usual care, waitlisted) or intervention group (6-week mind-body mobile application use). Randomization will be stratified on pain intensity and gender using computer generated block randomization to create varying block sizes of 4 and 8.
Masking Description: Participants in the control group will be aware that they have are serving as controls that have been wait-listed for access to the mobile application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mind-body mobile application (Experimental): Participants are asked to engage with a user-guided mobile application (app) that employs mind-based techniques that include: expressive writing, meditation, cognitive behavioural therapy, and pain education. The app also includes access to podcasts that focus on pain counselling and pain education.
  Interventions: Behavioral: Mind-body mobile application
- Control (No Intervention): Participants are asked to continue with usual care for pain treatments. They are asked not to start any new forms of treatment.

INTERVENTIONS:
Behavioral: Mind-body mobile application — Self-directed; Study team will recommend daily use of mobile app for 6 weeks with a minimum of 4 times/week usage of mobile app for 6 weeks. Frequency will be monitored via weekly surveys.
  Arms: Mind-body mobile application

SUMMARY:
We are investigating the effects of a mind-body based mobile application on the experience of chronic pain.

Participants meeting our criteria for chronic pain (confirmed via self-report) will complete an online baseline questionnaire. Eligible participants will be enrolled in the study and randomized into control (usual care, waitlisted) or intervention group (6-week mind-body based mobile application intervention). Randomization will be stratified by pain intensity and gender using computer-generated block randomization to create varying block sizes of 4 and 8. We will run the trial in multiple cohorts in series to obtain desired sample size.

All participants will complete online questionnaires at baseline and post-intervention at 6 weeks that measure pain intensity, interference with daily living, pain perceptions, mental health outcomes, and medication use. Participants will also complete weekly questionnaires on weeks 2 to 6 to gauge frequency of application usage (intervention) or other pain treatments (control). Participants in the intervention group will be asked to repeat the follow-up questionnaire at 12-weeks.

DETAILED DESCRIPTION:
See protocol for more details. (submitted at time of registration)

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 19 to 75 years with chronic pain.
* chronic pain is defined as having non-malignant chronic or persistent pain for at least 6 months.
* Participants must experience pain at least half the days in the last 6 months.
* Pain can include bodily pain or head (migraine) pain.

Exclusion Criteria:

* Individuals reporting a cognitive impairment that can interfere with completing questionnaires and using a mobile application.
* Individuals reporting any of the following psychiatric illness: schizophrenia, dissociative or personality disorders, bipolar disorder.
* Individuals reporting any of the following medical conditions: metastatic cancer, rheumatoid arthritis, lupus, scleroderma, polymyositis.
* Individuals reporting substance use disorder (within the last 6 months).
* Individuals that have previously used mind-body apps for the treatment of chronic pain.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia J Thomson, PhD, Principal Investigator — University of the Fraser Valley
Locations (1):
- University of the Fraser Valley, Chilliwack, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashar YK, Gordon A, Schubiner H, Uipi C, Knight K, Anderson Z, Carlisle J, Polisky L, Geuter S, Flood TF, Kragel PA, Dimidjian S, Lumley MA, Wager TD. Effect of Pain Reprocessing Therapy vs Placebo and Usual Care for Patients With Chronic Back Pain: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Jan 1;79(1):13-23. doi: 10.1001/jamapsychiatry.2021.2669. PMID 34586357
- [Background] Pfeifer AC, Uddin R, Schroder-Pfeifer P, Holl F, Swoboda W, Schiltenwolf M. Mobile Application-Based Interventions for Chronic Pain Patients: A Systematic Review and Meta-Analysis of Effectiveness. J Clin Med. 2020 Nov 5;9(11):3557. doi: 10.3390/jcm9113557. PMID 33167300
- [Background] Morone NE, Greco CM. Mind-body interventions for chronic pain in older adults: a structured review. Pain Med. 2007 May-Jun;8(4):359-75. doi: 10.1111/j.1526-4637.2007.00312.x. PMID 17610459
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. A classification of chronic pain for ICD-11. Pain. 2015 Jun;156(6):1003-1007. doi: 10.1097/j.pain.0000000000000160. No abstract available. PMID 25844555
- [Background] Borm GF, Fransen J, Lemmens WA. A simple sample size formula for analysis of covariance in randomized clinical trials. J Clin Epidemiol. 2007 Dec;60(12):1234-8. doi: 10.1016/j.jclinepi.2007.02.006. Epub 2007 Jun 6. PMID 17998077
- [Background] Schopflocher D, Taenzer P, Jovey R. The prevalence of chronic pain in Canada. Pain Res Manag. 2011 Nov-Dec;16(6):445-50. doi: 10.1155/2011/876306. PMID 22184555
- [Background] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Gatchel RJ, Peng YB, Peters ML, Fuchs PN, Turk DC. The biopsychosocial approach to chronic pain: scientific advances and future directions. Psychol Bull. 2007 Jul;133(4):581-624. doi: 10.1037/0033-2909.133.4.581. PMID 17592957
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Osman A, Barrios FX, Kopper BA, Hauptmann W, Jones J, O'Neill E. Factor structure, reliability, and validity of the Pain Catastrophizing Scale. J Behav Med. 1997 Dec;20(6):589-605. doi: 10.1023/a:1025570508954. PMID 9429990
- [Background] Kean J, Monahan PO, Kroenke K, Wu J, Yu Z, Stump TE, Krebs EE. Comparative Responsiveness of the PROMIS Pain Interference Short Forms, Brief Pain Inventory, PEG, and SF-36 Bodily Pain Subscale. Med Care. 2016 Apr;54(4):414-21. doi: 10.1097/MLR.0000000000000497. PMID 26807536

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three cohorts recruited in series for three study starts:
  Cohort 1: October 15 2021 Cohort 2: January 6 2022 Cohort 3: April 7 2022
  Randomized on October 15, 2022 (1); January 6, 2022 (2); and April 7, 2022.
Pre-assignment Details: Participants completed a baseline questionnaire following initial interest in the study. If the participants did not meet the criteria for chronic/persistent pain based on their responses to this survey, they were automatically excluded. If participants did not complete baseline (pre-randomization) survey such that primary outcome and randomization data was incomplete, they were excluded.
Period: Overall Study
Arm/Group | Mind-body Mobile Application | Control
Started | 98 | 100
Completed | 73 | 98
Not Completed | 25 | 2
Not completed — Lost to Follow-up | 10 | 2
Not completed — Withdrawal by Subject | 15 | 0

BASELINE CHARACTERISTICS:
Population: We report baseline characteristics for the full randomized sample (n = 198).
Groups:
- Total: Total of all reporting groups
Arm/Group | Mind-body Mobile Application | Control | Total
Number analyzed (Participants) | 98 | 100 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Missing age data for three participants in the intervention group, leaving n = 95 for mean age calculation.
  years
    number analyzed (Participants) | 95 | 100 | 195
    (all) | 46.6 (13.3) | 46.9 (13.0) | 46.7 (13.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Woman | 78 | 84 | 162
  Man | 15 | 14 | 29
  Non-binary | 3 | 2 | 5
  Prefer not to answer | 1 | 0 | 1
  Missing | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Population: Missing data on region of enrolment for 2 participants in the intervention group, leaving n = 96 for descriptive statistics for region.
  Participants
    Canada: number analyzed (Participants) | 96 | 100 | 196
    Canada | 86 | 90 | 176
    France: number analyzed (Participants) | 96 | 100 | 196
    France | 1 | 0 | 1
    United Kingdom: number analyzed (Participants) | 96 | 100 | 196
    United Kingdom | 2 | 0 | 2
    Israel: number analyzed (Participants) | 96 | 100 | 196
    Israel | 1 | 0 | 1
    Jamaica: number analyzed (Participants) | 96 | 100 | 196
    Jamaica | 1 | 0 | 1
    Trinidad and Tobago: number analyzed (Participants) | 96 | 100 | 196
    Trinidad and Tobago | 1 | 0 | 1
    United States: number analyzed (Participants) | 96 | 100 | 196
    United States | 4 | 8 | 12
    Greece: number analyzed (Participants) | 96 | 100 | 196
    Greece | 0 | 1 | 1
    Estonia: number analyzed (Participants) | 96 | 100 | 196
    Estonia | 0 | 1 | 1
Education [Count of Participants; unit: Participants] — Population: Missing data on education for n = 2 in intervention group and n = 2 in control group, leaving n = 96 intervention and n = 98 control.
  Participants
    High school or less: number analyzed (Participants) | 96 | 98 | 194
    High school or less | 13 | 10 | 23
    Trade or diploma: number analyzed (Participants) | 96 | 98 | 194
    Trade or diploma | 30 | 33 | 63
    Bachelor degree or higher: number analyzed (Participants) | 96 | 98 | 194
    Bachelor degree or higher | 53 | 55 | 108
Household income [Count of Participants; unit: Participants]
  < $34 999 | 29 | 27 | 56
  $35 000 to $49 999 | 12 | 3 | 15
  $50 000 to $74 999 | 16 | 20 | 36
  $75 000 to $99 999 | 13 | 20 | 33
  > $100 000 | 25 | 26 | 51
  Chose not to answer. | 3 | 4 | 7
Pain duration [Mean (Standard Deviation); unit: years] — Population: Missing data for 1 participant.
  years
    number analyzed (Participants) | 98 | 99 | 197
    (all) | 13.0 (11.0) | 14.2 (11.4) | 13.6 (11.2)
Diagnoses [Count of Participants; unit: Participants] — Diagnoses are not mutually exclusive as 24 participants had multiple diagnoses.
  Participants
    Fibromyalgia | 19 | 21 | 40
    Myalgic Encephalomyelitis | 4 | 6 | 10
    Osteoarthritis | 6 | 7 | 13
    Migraine | 10 | 13 | 23
    No formal diagnosis | 66 | 64 | 130
    Other (not including above conditions) | 11 | 7 | 18
Brief Pain Inventory (BPI) Pain Severity on average over past 24 hours [Mean (Standard Deviation); unit: units on a scale] — Single item scale within larger Brief Pain Inventory tool. Item scale ranges from 0 to 10. 0 = "no pain", 10 = "pain as bad as you can imagine". Higher scores indicate worse outcome, lower scores indicate better outcome.
  units on a scale | 5.5 (1.6) | 5.4 (1.5) | 5.45 (1.5)
Employment status [Count of Participants; unit: Participants]
  Employed (full or part time) | 50 | 47 | 97
  Retired | 10 | 13 | 23
  Other (student, homemaker) | 10 | 13 | 23
  Not able to work/on disability | 27 | 27 | 54
  Did not respond | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory-short Form (BPI-SF)
Description: Primary outcome of Pain Severity: Single item scale within larger Brief Pain Inventory tool. Item scale ranges from 0 to 10. 0 = "no pain", 10 = "pain as bad as you can imagine". Higher scores indicate worse outcome, lower scores indicate better outcome.
  Item range = (0,10).
  Primary outcome of Pain Interference: Item 9 on BPI measures interference with daily living. There are 7 items embedded within and each is scored on 11-point scales from 0 = "does not interfere" to 10 = "completely interferes" for interference with activities of daily living. Pain interference score is calculated as an average of the 7 items, with a range from 0 to 10. Higher scores represent worse outcomes.
Time Frame: Baseline, 6 weeks
Population: Intervention period was 6 weeks, and questionnaires were completed at baseline and at 6-weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mind-body Mobile Application | Control
Number analyzed (Participants) | 73 | 98
score on a scale
  BPI Average Pain Severity at baseline | 5.33 (1.47) | 5.35 (1.51)
  BPI Average Pain Severity at 6-weeks | 4.51 (1.74) | 5.16 (1.44)
  BPI Pain Interference at baseline | 5.97 (2.14) | 6.05 (2.26)
  BPI Pain interference at 6 weeks | 4.81 (2.32) | 5.49 (2.30)

2. Secondary Outcome: Patient Reported Outcome Measurement Information System (PROMIS) Short Form for Pain Intensity on Average
Description: Single item from PROMIS that measures self reported pain intensity on average over 7 days.
  5-point scale: 1 = "had no pain" to 5 = "very severe pain" Scale range = (1,5). Higher score indicates worse outcome.
Time Frame: baseline, 6 weeks
Population: Missing PROMIS intensity data for one participant in the control group at 6 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mind-body Mobile Application | Control
Number analyzed (Participants) | 73 | 97
units on a scale
  PROMIS Pain Intensity on average at baseline | 2.99 (0.59) | 3.22 (0.60)
  PROMIS Pain Intensity on average at 6-weeks | 2.81 (0.54) | 3.08 (0.61)

3. Secondary Outcome: Patient Reported Outcome Measurement Information System (PROMIS) Short Form 8a Pain Interference
Description: Measures self reported pain interference in daily activities (over 7 days). 8 items are added together for a sum score.
  Each item uses 5-pt Likert scale from 1 = "not at all" to 5 = "very much" (regarding pain interference).
  Scale range = 8 to 40. Higher scores indicate worse outcomes.
Time Frame: baseline, 6 weeks
Population: Missing PROMIS data for one participant in the control group at 6 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mind-body Mobile Application | Control
Number analyzed (Participants) | 73 | 97
score on a scale
  Total PROMIS Pain Interference at baseline | 28.22 (7.30) | 29.01 (7.46)
  Total PROMIS Pain Interference at 6-weeks | 16.71 (8.36) | 19.63 (8.28)

4. Secondary Outcome: Pain Catastrophizing Questionnaire (PCS)
Description: Measures thoughts and perceptions of pain, 13 items, scored using 5-pt Likert scale 0 = "not at all" to 4 = "all the time".
  Scores are the sum of all items. min score = 0; max score = 52. Higher scores indicate worse outcomes.
Time Frame: baseline, 6 weeks
Population: Missing PCS data for one participant in the control group at 6 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mind-body Mobile Application | Control
Number analyzed (Participants) | 73 | 97
score on a scale
  Total PCS Scores at baseline | 22.55 (12.22) | 23.13 (11.30)
  Total PCS Scores at 6-weeks | 15.92 (11.48) | 20.38 (12.0)

5. Secondary Outcome: DASS-21 (Depression, Anxiety, and Stress Scale)
Description: Measures self reported emotional states, three subscales: depression, anxiety, stress (each 7 items) Items scored on 4-point Likert scale: 0 = "did not apply to me at all" to 3 = "applied to me very much or most of the time".
  Scores for each subscale are summed. Scores are then multiplied by 2 to calculate final score for each subscale.
  Scale ranges for each subscale is from 0 to 42 (after doubling of scores). Higher scores indicate worse outcomes.
Time Frame: baseline, 6 weeks
Population: Missing depression data for two participants in the control group. Missing anxiety data for one participant in the intervention group and two participants in the control group.
  Missing stress data for two participants in the intervention group and two participants in the control group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mind-body Mobile Application | Control
Number analyzed (Participants) | 73 | 96
score on a scale
  Total Depression Score at baseline | 14.57 (9.52) | 14.52 (9.84)
  Total Depression Score at 6-weeks | 11.97 (9.09) | 14.85 (10.75)
  Total Anxiety Score at baseline: number analyzed (Participants) | 72 | 96
  Total Anxiety Score at baseline | 9.89 (7.85) | 8.92 (7.13)
  Total Anxiety Score at 6-weeks: number analyzed (Participants) | 72 | 96
  Total Anxiety Score at 6-weeks | 7.31 (7.73) | 9.46 (7.74)
  Total Stress Score at baseline: number analyzed (Participants) | 71 | 96
  Total Stress Score at baseline | 16.54 (8.78) | 15.35 (8.33)
  Total Stress Score at 6-weeks: number analyzed (Participants) | 71 | 96
  Total Stress Score at 6-weeks | 13.63 (8.14) | 15.46 (8.63)

6. Secondary Outcome: Quality of Life Short Form 12 (SF-12) Physical (PCS-12) and Mental (MCS-12) Component Summary Scores (Z-scores; Normalized Based on US General Population)
Description: Measures self-reported impact of health on daily life. The SF-12 is a brief version of the longer SF-36 and contains 12 items measured using a variety of Likert scales and dichotomous yes/no scales, with each item response assigned a numerical weight.
  PCS and MCS are component z-scores that are calculated using regression weights and constants for each (mental and physical) which have been derived from a U.S. population.
  Each item response choice category is coded as an indicator variable (scored 1 / 0). Indicator variables are weighted using regression coefficients from the US population for the MCS and PCS. The weighted scores across all items are then summed and are added to a constant (regression intercept) to obtain summary scores. Score ranges 0 to 100. Normalized score such that component scales have a mean of 50 and standard deviation of 10 in the general population.
  Lower scores indicate worse outcomes. Higher scores indicate better
Time Frame: baseline, 6 weeks
Population: Missing Physical Component Score data for three participants in the control group.
  Missing Mental Component Score data for three participants in the control group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mind-body Mobile Application | Control
Number analyzed (Participants) | 73 | 95
score on a scale
  QOL Physical Component Score at baseline | 25.21 (11.07) | 21.60 (9.58)
  QOL Physical Component Score at 6-weeks | 29.27 (11.37) | 23.89 (11.36)
  QOL Mental Component Score at baseline | 47.83 (5.47) | 49.18 (6.74)
  QOL Mental Component Score at 6-weeks | 49.22 (6.39) | 50.05 (6.97)

7. Secondary Outcome: Brief Pain Inventory-short Form (BPI-SF)
Description: Measures self reported pain severity; Pain interference (over past 24 hours) Only measured in the intervention group (as wait-listed controls had accessed the mobile app and were released from the study).
  BPI Pain Severity: single item scale within larger Brief Pain Inventory tool. Item scale ranges from 0 to 10. 0 = "no pain", 10 = "pain as bad as you can imagine". Higher scores indicate worse outcome, lower scores indicate better outcome.
  Item range = (0,10).
  BPI Pain Interference: Item 9 on BPI measures interference with daily living. There are 7 items embedded within and each is scored on 11-point scales from 0 = "does not interfere" to 10 = "completely interferes" for interference with activities of daily living. Pain interference score is calculated as an average of the 7 items, with a range from 0 to 10. Higher scores represent worse outcomes.
Time Frame: 12 weeks
Population: Members of the intervention group who completed the additional 12 week follow up (intervention ended at 6 weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Mind-body Mobile Application: Participants in the intervention group completed an additional follow-up survey at 12 weeks. There was no requirement to continue using the mobile app, but we collected data on who continued using the app.
Arm/Group | Mind-body Mobile Application
Number analyzed (Participants) | 65
score on a scale
  BPI Pain intensity on average (24 hours) | 4.60 (1.70)
  Pain interference (24 hours) | 4.85 (2.49)

8. Secondary Outcome: PROMIS Pain Intensity Short Form
Description: as for outcome 2
Time Frame: 12 weeks
Population: Members of the intervention group who completed the additional 12 week follow up (intervention ended at 6 weeks).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mind-body Mobile Application
Number analyzed (Participants) | 65
units on a scale | 2.74 (0.54)

9. Secondary Outcome: Medication Use
Description: Self-reported quantify of medication use (number of participant reporting regular usage).
  Note: this was a change from original plan for reporting. We have only reported frequencies of use (generally), and omitted details regarding dosage and number of pills as it was decided that this was beyond the scope of our team and trial. We also did not compare baseline to 6 weeks for the same reason.
Time Frame: 6 weeks
Population: Medication categories are not mutually exclusive as many report usage of multiple classes of drugs.
Measure: Number; unit: participants
Arm/Group | Mind-body Mobile Application | Control
Number analyzed (Participants) | 73 | 98
participants
  Non-opioid analgesics | 48 | 59
  Opioid analgesics | 11 | 29
  Anti-depressants (SSRI, SSNI, TCA) | 20 | 27
  Anti-convulsants | 13 | 31
  Anti-spasmodics | 8 | 9
  Cannabanoids | 6 | 10
  CNS depressants | 5 | 8
  Other medicines related to pain | 9 | 5

10. Secondary Outcome: PROMIS Pain Interference Short Form 8a
Description: as for outcome 3
Time Frame: 12 weeks
Population: Members of the intervention group who completed the additional 12 week follow up (intervention ended at 6 weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mind-body Mobile Application
Number analyzed (Participants) | 65
score on a scale | 24.34 (7.54)

11. Secondary Outcome: Pain Catastrophizing Questionnaire (PCS)
Description: as for outcome 4
Time Frame: 12 weeks
Population: Members of the intervention group who completed the additional 12 week follow up (intervention ended at 6 weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mind-body Mobile Application
Number analyzed (Participants) | 65
score on a scale | 16.46 (12.83)

12. Secondary Outcome: Quality of Life Short Form 12 (SF-12) Physical (PCS-12) and Mental (MCS-12) Component Summary Scores (Z-scores; Normalized Based on US General Population)
Description: Measures self-reported impact of health on daily life. The SF-12 is a brief version of the longer SF-36 and contains 12 items measured using a variety of Likert scales and dichotomous yes/no scales, with each item response assigned a numerical weight.
  PCS and MCS are component z-scores that are calculated using regression weights and constants for each (mental and physical) which have been derived from a U.S. population.
  Each item response choice category is coded as an indicator variable (scored 1 / 0). Indicator variables are weighted using regression coefficients from the US population for the MCS and PCS. The weighted scores across all items are then summed and are added to a constant (regression intercept) to obtain summary scores. Score ranges 0 to 100. Normalized score such that component scales have a mean of 50 and standard deviation of 10 in the general population.
  Lower scores indicate worse outcomes. Higher scores indicate better outcomes.
Time Frame: 12 weeks
Population: Members of the intervention group who completed the additional 12 week follow up (intervention ended at 6 weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mind-body Mobile Application
Number analyzed (Participants) | 65
score on a scale
  Physical Component Score (SF12) at 12 weeks | 27.66 (10.34)
  Mental Component Score (SF12) at 12 weeks | 50.20 (7.63)

13. Secondary Outcome: DASS-21 (Depression, Anxiety, Stress Scale - 21 Items)
Description: as for outcome 5
Time Frame: 12 weeks
Population: See above 12 week data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mind-body Mobile Application
Number analyzed (Participants) | 65
score on a scale
  Depression | 6.32 (4.99)
  Anxiety: number analyzed (Participants) | 64
  Anxiety | 4.20 (3.72)
  Stress: number analyzed (Participants) | 64
  Stress | 7.58 (4.71)

ADVERSE EVENTS:
Time Frame: 6 weeks.
Description: There were no adverse events reported at the 6-week follow up. We have data for completed cases (n = 73 intervention, n = 98 control. There was an open ended question to report anything not captured by our survey. No participants reported any adverse events due to the intervention. We do not have data for those that were lost to follow up.
  Only the intervention group was followed at 12 weeks. No adverse events reported in the intervention group at 12 weeks (n = 65 completed survey).
Arm/Group | Mind-body Mobile Application | Control
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/98
Other Adverse Events (participants affected / at risk) | 0/73 | 0/98

LIMITATIONS AND CAVEATS:
Note the data reported here are for complete cases (n = 171) and represent means from raw data (not estimated means). n = 73 intervention, n = 98 usual care (with missing data in secondary outcomes noted). Formal analysis presented in reports include intention to treat sample (n = 198) and estimated marginal means are reported elsewhere.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT05090683/Prot_SAP_000.pdf